CLINICAL TRIAL: NCT05262244
Title: Targeted Fluorescence Imaging Using Bevacizumab-800CW Within Age-related Macular Degeneration (AMD) Patients to Evaluate the Upregulation of VEGF
Brief Title: Targeted Fluorescence Imaging in AMD
Acronym: LEAF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL78391.056.21
Record Dates: First submitted 2021-11-19; First posted 2022-03-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-03

CONDITIONS: Age-Related Macular Degeneration; NAMD
Keywords: fluorescence, ophthalmology, bevacizumab-800CW, nAMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: First a dose finding study is performed using bevacizumab-800CW within the AMD patient group. Using the optimal dose and if fluorescence is visible, additional inclusion of patients with the optimal dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AMD with bevacizumab-800CW (Experimental): Patients with AMD receive bevacizumab-800CW followed by angiography
  Interventions: Drug: Bevacizumab-IRDye800CW

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — Bevacizumab-800CW is administered to the patient and angiography is performed before and directly after tracer administration and after 48-96 hours.

SUMMARY:
Rationale:

To track performance of intravitreal distribution of anti-VEGF-A (Bevazicumab-800CW) and provide information about neovascularization and inflammation in Age-Related Macular Degeneration (AMD), thereby predicting progression and optimizing treatment

Objective:

To determine the safety and feasibility of fluorescence imaging of the eye with the fluorescent tracer bevacizumab-800CW for identification AMD with scanning laser angiography

Study design:

A non-randomized, non-blinded, prospective, single-center feasibility study.

Study population:

Patients group: patients with naïve wet AMD and wet AMD aged >60 years old with current treatment of anti-VEGF intravitreal.

Control group: patients with naïve wet AMD and wet AMD aged >60 years old with current treatment of anti-VEGF intravitreal

Intervention (if applicable):

Intravenous injection of bevacizumab-800CW in the patient group.

Main study parameters/endpoints:

Safety and feasibility of the intravenous tracer bevacizumab-800CW in patients with naïve wet AMD and wet AMD by observing the uptake in retinal, choroid and neovascular tissue.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: No risk described in other (running) studies on intravenous injection with bevacizumab-800 CW. Patients need to come back 48-96 hours after injection and the eye measurements take about half an hour longer.

There is no benefit with participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either naïve wet AMD or wet AMD receiving standard care of anti-VEGF therapy
* Aged >60 years old

Optional: Patients already included in fluorescence study which involves Bevacizumab-800CW

Exclusion Criteria:

* Eye pathology interfering with retinal imaging;
* Patients with psychological diseases or medical issues who are not able to sign informed consent form;
* Concurrent uncontrolled medical conditions;
* Received a different investigational drug within 30 days prior to the dose of bevacizumab-800CW;
* History of infusion reactions to bevacizumab or other monoclonal antibody.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Safety: number of participants with symptoms or changes in vital signs (blood pressure, heart rate and temperature) that are related to administration of bevacizumab-800CW | Directly after administration until 96 hours after.
  To determine the safety of bevacizumab-800CW in patients with AMD by monitoring of vital signs (blood pressure, heart rate and temperature), before and until one hour after administration.
Feasibility: the possibility of measuring the specific uptake of fluorescence within the eye using both scanning laser angiography and optical coherence tomography. | Directly after administration until 96 hours after
  The target-to-background radio will be measured during fluorescence imaging and compared with imaging before tracer administration.

SECONDARY OUTCOMES:
Determination of the most optimal dose of bevacizumab-800CW for fluorescence imaging of the eye vascularization. | Directly after administration until 96 hours after.
  The target-to-background radio will be calculated and the dose with the highest ratio will be used as most optimal dose.
Correlation of the fluorescence intensity, target-to-background ratio (TBR), with disease identification | Up to 1 year
  The target-to-background ratio will be calculated and compared to the disease identification scale.
Correlation between fluorescence intensity and clinical score | Up to 1 year
  The subtype and severity of neovascularization will be determined and used as a clinical score.
Correlation of VEGF expression within the tear fluid with the fluorescent signal | Up to 1 year
  Gather tear fluid with Schirmer strips and using ELISA to extract the VEGF concentration and correlate this with the fluorescence signal

CONTACTS AND LOCATIONS:
Overall Officials: W. B Nagengast, MD, PhD, PharmD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University medical center Groningen (UMCG), Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No